CLINICAL TRIAL: NCT03502070
Title: A Multicenter, Human Factors Validation Study in Cystic Fibrosis Patients Aged 6 Years and Older to Evaluate the User Interface of TOBI® Podhaler™ (Tobramycin Inhalation Powder) Using Placebo Capsules
Brief Title: Human Factors Study to Validate the User Interface of TOBI Podhaler Using Placebo Capsules
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mylan Inc. (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CTBM100C2419
Record Dates: First submitted 2018-03-29; First posted 2018-04-18 (Actual); Results first posted 2020-06-30 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Cystic Fibrosis
Keywords: CF, Human Factors, TOBI® Podhaler™, user interface, IFU
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Open-Label Placebo (Other): One dose (4 capsules) of placebo
  Interventions: Drug: Placebo; Device: Tobi Podhaler

INTERVENTIONS:
Drug: Placebo — One dose (4 capsules) of placebo
Device: Tobi Podhaler — The placebo capsule has to be released from the blister card and inserted into the Podhaler device. The device is then actuated and the study drug is inhaled according to the instructions for use

SUMMARY:
The purpose of this study is to validate the user interface of TOBI Podhaler by establishing that the product can support safe and effective use for the intended users

DETAILED DESCRIPTION:
The objective is to conduct a human factors validation study to demonstrate that the user interface of TOBI® Podhaler™ can support safe and effective use for the intended users. The human factors validation study will be conducted in patients with cystic fibrosis aged 6 years and older under simulated yet representative of realistic use conditions where patients with no prior training or use of TOBI® Podhaler™ will be asked to inhale the contents of placebo capsules through the Podhaler device. Due to the use of placebo capsules, the study is considered an interventional clinical study and will be conducted accordingly. The study is an open label, un-blinded, non-randomized study which consists of one visit.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent or, parent/guardian consent and where applicable pediatric assent, must be obtained before any assessment is performed
* Male and female subjects aged 6 years and older
* Confirmed diagnosis of CF by one or more of the following tests for CF as documented in the patient's medical history : (1) quantitative pilocarpine iontophoresis sweat chloride test of > 60 mmol/L or 60 mEq/L, (2) genotype with identifiable CF-causing mutations on both chromosomes, (3) an abnormal nasal transepithelial potential difference characteristic of CF
* FEV1 value must be at least 25% of normal predicted values for age, sex, and height as documented in the patient's medical history (historical values within 3 months can be used for this criterion).
* Able to comply with all protocol requirements
* Clinically stable in the opinion of the investigator

Exclusion Criteria:

* Subjects currently enrolled in studies that are not considered as observational non-investigational studies
* Subjects or caregivers who have used the Podhaler device previously
* Hemoptysis more than approximately 60 mL at any time within 30 days prior to enrollment
* History of hypersensitivity to the inhaled placebo dry powder (DSPC and/or calcium chloride powder)
* Signs and symptoms of acute pulmonary disease, e.g. pneumonia, pneumothorax, bronchospasm, acute respiratory infection
* Clinically significant conditions or findings at enrollment that might interfere with the accurate and valid assessment of this study
* Subjects or caregivers who are considered potentially unreliable or considered unlikely to be compliant within the trial
* Pregnant women

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2019-06-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Batchelor Childrens Research Institute, Miami, Florida
  - University of Miami Hospital, Miami, Florida
  - Nemours Childrens Hospital, Orlando, Florida
  - Nemour's Children's Clinic - Pensacola, Pensacola, Florida
  - Tulane Lakeside Hospital for Women and Children, New Orleans, Louisiana
  - Toledo Childrens Hospital, Toledo, Ohio
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Respiratory Diseases of Children and Adolescents, Oklahoma City, Oklahoma
  - VCU Children's Pavilion, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open-Label Placebo
Started | 47
Completed | 45
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Screen Failure | 1

BASELINE CHARACTERISTICS:
Arm/Group | Open-Label Placebo
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.5 (12.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 41
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Critical Use Errors and Close Calls Associated With the Simulated Inhalation of One Dose Using TOBI Podhaler
Description: Critical use errors and close calls for the following: placing of capsule into the top of the mouthpiece, failure to replace mouthpiece, failure to adequately pierce capsule, failure to release before inhaling, multiple piercing of capsule, exhalation into mouthpiece, inadequate seal around mouthpiece, inadequate inhalation technique, failure to use reserve device when capsule not adequately pierced, failure to administer 4 capsules per dose, swallowing of capsule
Time Frame: 1 Day
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Placebo
Number analyzed (Participants) | 45
Participants | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of signing Informed Consent through completion of their study visit, 1 day
Arm/Group | Open-Label Placebo
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 1/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label Placebo (N=45)
Subject Accidentally Kicked Himself Causing A Wart To Bleed On His Leg (Injury, poisoning and procedural complications) | 1 (1)
Wart On Leg (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Wart Bleed On Leg (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-11-12): https://cdn.clinicaltrials.gov/large-docs/70/NCT03502070/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-04): https://cdn.clinicaltrials.gov/large-docs/70/NCT03502070/SAP_001.pdf